CLINICAL TRIAL: NCT02029872
Title: Stop Community MRSA Colonization Among Patients (SUSTAIN)
Brief Title: Stop Community MRSA Colonization Among Patients
Acronym: SUSTAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00079147
Record Dates: First submitted 2013-12-18; First posted 2014-01-08 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: MRSA
Keywords: MRSA; colonization; decolonization
MeSH Terms: interventions — chlorhexidine gluconate; Chlorhexidine; Mupirocin; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual plus household (Active Comparator): Standard decolonization regimen for individual plus household: 7 day course of nasal mupirocin calcium 2% ointment applied inside the nose twice daily 4% chlorhexidine gluconate (soap) used in the shower/bath every day for 7 days. For individuals colonized within the throat we will add chlorhexidine gluconate oral rinse 0.12% used in a gargle and spit fashion twice daily for 7 days.
  Interventions: Drug: Chlorhexidine gluconate soap; Drug: Chlorhexidine gluconate oral rinse; Drug: Mupirocin calcium 2 % ointment
- Individual alone (Active Comparator): Standard decolonization regimen for the individual alone: 7 day course of nasal mupirocin calcium 2% ointment applied inside the nose twice daily, plus a 4% chlorhexidine gluconate (soap) used in the shower/bath every day for 7 days. For individuals colonized within the throat we will add chlorhexidine gluconate oral rinse 0.12% used in a gargle and spit fashion twice daily for 7 days.
  Interventions: Drug: Chlorhexidine gluconate soap; Drug: Chlorhexidine gluconate oral rinse; Drug: Mupirocin calcium 2 % ointment

INTERVENTIONS:
Drug: Chlorhexidine gluconate soap — 4% chlorhexidine gluconate (soap)
  Other Names: Hibiclens
Drug: Chlorhexidine gluconate oral rinse — chlorhexidine gluconate oral rinse 0.12%
  Other Names: Chlorhexidine
Drug: Mupirocin calcium 2 % ointment — nasal mupirocin calcium 2% ointment
  Other Names: Mupirocin

SUMMARY:
This research is being done to learn more about an approach to remove Methicillin resistant Staphylococcus aureus (MRSA) in patients who are carriers of the bacteria in outpatient settings and among their household members and sexual partners.

MRSA is a type of bacteria or germ that can cause bad infections of the skin that can make people very sick. The bacteria have been seen in a high number of persons in the Baltimore area and in hospitals throughout the country. MRSA can be spread from person to person, particularly in homes and among family members and sexual partners.

There are three things the investigators hope to learn from this research study:

First, the investigators want to find a way to prevent MRSA infections in outpatient settings. By asking questions, the investigators want to look at the things that may increase the risk of having this type of bacteria in you and your family members.

Second, the investigators have soaps and oral rinses (Chlorhexidine) and medications (antibiotics; Mupirocin ointment) that have been shown to be effective at removing MRSA. The investigators want to determine if these antibiotics and soaps are best used for everyone in the household or only the individual with known MRSA.

Third, as the investigators, we want to learn more about the bacteria by looking at it on the inside. The investigators will do laboratory tests on samples we collect, to learn how MRSA bacteria grow, reproduce and how it develops to behave differently than other types of MRSA bacteria.

DETAILED DESCRIPTION:
Methicillin resistant Staphylococcus aureus (MRSA) kills more patients in the United States (U.S.) than Acquired Immunodeficiency Syndrome (AIDS). Further, persons living with Human Immunodeficiency Virus (HIV) experience MRSA infection at significantly higher rates than the general population (12.3/ 1000 person years compared to 1 to 2/1000 person years) and MRSA remains a substantial reason for hospital admission among this patient population. Colonization with Staphylococcus aureus is a major risk factor for infection in persons living with HIV and AIDS (PLWHA) and eradication of MRSA colonization reduces the occurrence of subsequent infection in patients. Household contacts with MRSA colonization increase failure rates of decolonization. The clinical practice guidelines for MRSA management from the Infectious Diseases Society of America (IDSA) recommend providing decolonization to persons with repeated skin and soft tissue infections as well as their household contacts; however, the guidelines report that evidence is limited in support of this recommendation. Additionally, these recommendations do not include sexual partners outside the home and there is mounting evidence of MRSA transmission between sexual partners and sexual networks. Strategies that reduce the spread of MRSA among people living with HIV/AIDS (PLWHA) are vitally needed to reduce this disparity.

To assess colonization prevalence among PLWHA, investigators conducted an epidemiologic evaluation of MRSA among persons within the Johns Hopkins University AIDS Service (JHUAS). The study included 500 subjects (65.8 % male) along with the sexual partners of 35 subjects. The MRSA colonization prevalence was 16.8% among subjects and 37% (17/35) in their sexual partners (unpublished data). These findings demonstrate an exceptional difference in colonization prevalence in PLWHA compared to the US population and supports the need for further research to understand decolonization regimens that evaluate outcomes for individual decolonization only compared to the inclusion household and/or sexual partner interventions. We propose a randomized controlled trial (RCT) among 100 PLWHA (50 per arm) within the JHUAS to evaluate an individual versus household/sexual partner decolonization intervention.

The specific aims of the proposed RCT are:

1. To compare a MRSA decolonization protocol for the colonized individual (index) versus the index plus their household member and/or routine sexual partner(s).

   H0: Index plus household/sexual partner(s) decolonization will be associated with a lower occurrence of MRSA colonization at 6 months after completion of decolonization protocol.
2. To estimate the intervention effect size and develop an intervention fidelity assessment plan to scale the intervention into a larger multi-city R01 application.
3. To determine the molecular characteristics and antimicrobial susceptibilities of both the clinical and colonizing isolates among index patient as well as household members.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, 21 years of age and older, of all racial and ethnic groups, receiving care within the Johns Hopkins University AIDS Service who have a prior history of MRSA colonization are eligible to participate as the index HIV positive subject
* have at least two members in the household and/or a sexual partner
* subjects must be willing to be randomized to either arm of the study, including randomization to household and/or sexual partner evaluation that includes home visits
* Sexual partners and/or household members will also be required to provide informed consent
* Subjects and their contacts must have no documented or reported allergies to any agent used in the standardized decolonization regimen
* Parental assent will be required for household members less than 7 years of age

Exclusion Criteria:

* individuals who live alone and have no active sexual partners
* allergy to any component of decolonization protocol
* individuals who are unable to provide written informed consent

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Farley, PhD, MPH, NP, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klevens RM, Morrison MA, Nadle J, Petit S, Gershman K, Ray S, Harrison LH, Lynfield R, Dumyati G, Townes JM, Craig AS, Zell ER, Fosheim GE, McDougal LK, Carey RB, Fridkin SK; Active Bacterial Core surveillance (ABCs) MRSA Investigators. Invasive methicillin-resistant Staphylococcus aureus infections in the United States. JAMA. 2007 Oct 17;298(15):1763-71. doi: 10.1001/jama.298.15.1763. PMID 17940231
- [Background] Crum-Cianflone N, Weekes J, Bavaro M. Recurrent community-associated methicillin-resistant Staphylococcus aureus infections among HIV-infected persons: incidence and risk factors. AIDS Patient Care STDS. 2009 Jul;23(7):499-502. doi: 10.1089/apc.2008.0240. PMID 19530952
- [Background] Crum-Cianflone NF, Grandits G, Echols S, Ganesan A, Landrum M, Weintrob A, Barthel R, Agan B; Infectious Disease Clinical Research Program. Trends and causes of hospitalizations among HIV-infected persons during the late HAART era: what is the impact of CD4 counts and HAART use? J Acquir Immune Defic Syndr. 2010 Jul;54(3):248-57. doi: 10.1097/qai.0b013e3181c8ef22. PMID 20658748
- [Background] Shet A, Mathema B, Mediavilla JR, Kishii K, Mehandru S, Jeane-Pierre P, Laroche M, Willey BM, Kreiswirth N, Markowitz M, Kreiswirth BN. Colonization and subsequent skin and soft tissue infection due to methicillin-resistant Staphylococcus aureus in a cohort of otherwise healthy adults infected with HIV type 1. J Infect Dis. 2009 Jul 1;200(1):88-93. doi: 10.1086/599315. PMID 19463064
- [Background] Buehlmann M, Frei R, Fenner L, Dangel M, Fluckiger U, Widmer AF. Highly effective regimen for decolonization of methicillin-resistant Staphylococcus aureus carriers. Infect Control Hosp Epidemiol. 2008 Jun;29(6):510-6. doi: 10.1086/588201. PMID 18510460
- [Background] Ammerlaan HS, Kluytmans JA, Berkhout H, Buiting A, de Brauwer EI, van den Broek PJ, van Gelderen P, Leenders SA, Ott A, Richter C, Spanjaard L, Spijkerman IJ, van Tiel FH, Voorn GP, Wulf MW, van Zeijl J, Troelstra A, Bonten MJ; MRSA Eradication Study Group. Eradication of carriage with methicillin-resistant Staphylococcus aureus: determinants of treatment failure. J Antimicrob Chemother. 2011 Oct;66(10):2418-24. doi: 10.1093/jac/dkr250. Epub 2011 Jun 30. PMID 21719471
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF; Infectious Diseases Society of America. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis. 2011 Feb 1;52(3):e18-55. doi: 10.1093/cid/ciq146. Epub 2011 Jan 4. PMID 21208910
- [Background] Crum-Cianflone NF, Shadyab AH, Weintrob A, Hospenthal DR, Lalani T, Collins G, Mask A, Mende K, Brodine SK, Agan BK; Infectious Disease Clinical Research Program HIV Working Group. Association of methicillin-resistant Staphylococcus aureus (MRSA) colonization with high-risk sexual behaviors in persons infected with human immunodeficiency virus (HIV). Medicine (Baltimore). 2011 Nov;90(6):379-389. doi: 10.1097/MD.0b013e318238dc2c. PMID 22033452
- [Background] Shadyab AH, Crum-Cianflone NF. Methicillin-resistant Staphylococcus aureus (MRSA) infections among HIV-infected persons in the era of highly active antiretroviral therapy: a review of the literature. HIV Med. 2012 Jul;13(6):319-32. doi: 10.1111/j.1468-1293.2011.00978.x. Epub 2012 Jan 25. PMID 22276696
- [Background] Graham PL 3rd, Lin SX, Larson EL. A U.S. population-based survey of Staphylococcus aureus colonization. Ann Intern Med. 2006 Mar 7;144(5):318-25. doi: 10.7326/0003-4819-144-5-200603070-00006. PMID 16520472
- [Background] Diep BA, Chambers HF, Graber CJ, Szumowski JD, Miller LG, Han LL, Chen JH, Lin F, Lin J, Phan TH, Carleton HA, McDougal LK, Tenover FC, Cohen DE, Mayer KH, Sensabaugh GF, Perdreau-Remington F. Emergence of multidrug-resistant, community-associated, methicillin-resistant Staphylococcus aureus clone USA300 in men who have sex with men. Ann Intern Med. 2008 Feb 19;148(4):249-57. doi: 10.7326/0003-4819-148-4-200802190-00204. Epub 2008 Jan 30. PMID 18283202
- [Background] Crum-Cianflone NF, Burgi AA, Hale BR. Increasing rates of community-acquired methicillin-resistant Staphylococcus aureus infections among HIV-infected persons. Int J STD AIDS. 2007 Aug;18(8):521-6. doi: 10.1258/095646207781439702. PMID 17686212
- [Background] Skiest DJ, Brown K, Cooper TW, Hoffman-Roberts H, Mussa HR, Elliott AC. Prospective comparison of methicillin-susceptible and methicillin-resistant community-associated Staphylococcus aureus infections in hospitalized patients. J Infect. 2007 May;54(5):427-34. doi: 10.1016/j.jinf.2006.09.012. Epub 2006 Oct 27. PMID 17070598
- [Background] Al-Rawahi GN, Schreader AG, Porter SD, Roscoe DL, Gustafson R, Bryce EA. Methicillin-resistant Staphylococcus aureus nasal carriage among injection drug users: six years later. J Clin Microbiol. 2008 Feb;46(2):477-9. doi: 10.1128/JCM.01596-07. Epub 2007 Nov 26. PMID 18039800
- [Background] Huang H, Cohen SH, King JH, Monchaud C, Nguyen H, Flynn NM. Injecting drug use and community-associated methicillin-resistant Staphylococcus aureus infection. Diagn Microbiol Infect Dis. 2008 Apr;60(4):347-50. doi: 10.1016/j.diagmicrobio.2007.11.001. Epub 2008 Feb 21. PMID 18178362
- [Background] Lee NE, Taylor MM, Bancroft E, Ruane PJ, Morgan M, McCoy L, Simon PA. Risk factors for community-associated methicillin-resistant Staphylococcus aureus skin infections among HIV-positive men who have sex with men. Clin Infect Dis. 2005 May 15;40(10):1529-34. doi: 10.1086/429827. Epub 2005 Apr 13. PMID 15844078
- [Background] Mathews WC, Caperna JC, Barber RE, Torriani FJ, Miller LG, May S, McCutchan JA. Incidence of and risk factors for clinically significant methicillin-resistant Staphylococcus aureus infection in a cohort of HIV-infected adults. J Acquir Immune Defic Syndr. 2005 Oct 1;40(2):155-60. doi: 10.1097/01.qai.0000179464.40948.b9. PMID 16186732
- [Background] Drapeau CM, Angeletti C, Festa A, Petrosillo N. Role of previous hospitalization in clinically-significant MRSA infection among HIV-infected inpatients: results of a case-control study. BMC Infect Dis. 2007 Apr 30;7:36. doi: 10.1186/1471-2334-7-36. PMID 17470274
- [Background] Fritz SA, Hogan PG, Hayek G, Eisenstein KA, Rodriguez M, Epplin EK, Garbutt J, Fraser VJ. Household versus individual approaches to eradication of community-associated Staphylococcus aureus in children: a randomized trial. Clin Infect Dis. 2012 Mar;54(6):743-51. doi: 10.1093/cid/cir919. Epub 2011 Dec 23. PMID 22198793
- [Background] Ammerlaan HS, Kluytmans JA, Berkhout H, Buiting A, de Brauwer EI, van den Broek PJ, van Gelderen P, Leenders SA, Ott A, Richter C, Spanjaard L, Spijkerman IJ, van Tiel FH, Voorn GP, Wulf MW, van Zeijl J, Troelstra A, Bonten MJ; MRSA Eradication Study Group. Eradication of carriage with methicillin-resistant Staphylococcus aureus: effectiveness of a national guideline. J Antimicrob Chemother. 2011 Oct;66(10):2409-17. doi: 10.1093/jac/dkr243. Epub 2011 Jun 30. PMID 21719473
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Farley JE, Stamper PD, Ross T, Cai M, Speser S, Carroll KC. Comparison of the BD GeneOhm methicillin-resistant Staphylococcus aureus (MRSA) PCR assay to culture by use of BBL CHROMagar MRSA for detection of MRSA in nasal surveillance cultures from an at-risk community population. J Clin Microbiol. 2008 Feb;46(2):743-6. doi: 10.1128/JCM.02071-07. Epub 2007 Dec 5. PMID 18057129
- [Background] Farley JE, Ross T, Stamper P, Baucom S, Larson E, Carroll KC. Prevalence, risk factors, and molecular epidemiology of methicillin-resistant Staphylococcus aureus among newly arrested men in Baltimore, Maryland. Am J Infect Control. 2008 Nov;36(9):644-50. doi: 10.1016/j.ajic.2008.05.005. Epub 2008 Oct 3. PMID 18834755

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from January 2014-March 2015 in an outpatient HIV clinic in Baltimore, Maryland
Pre-assignment Details: Enrolled participants were screened for Methicillin-resistant Staphylococcus aureus (MRSA). Only those with a positive MRSA swab in any body site (nares, throat, perineum, rectum, vagina) were randomized to an arm of the study to receive the decolonization protocol.
Period: Overall Study
Arm/Group | Individual Alone | Individual Plus Household
Started | 9 | 9
Completed | 7 | 6
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: 77 enrolled participants were screened for MRSA. Only those with a positive MRSA swab in any body site (nares, throat, perineum, rectum, vagina) were randomized to an arm of the study to receive the decolonization protocol. 59 participants were not randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Alone | Individual Plus Household | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (4.2) | 51.4 (12.2) | 50.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 2 | 1 | 3
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18
Cluster of Differentiation 4 (CD4) T-cell count [Mean (Standard Deviation); unit: cells/mm^3] — CD4 cells per cubic millimeter of blood
  cells/mm^3 | 676 (451) | 687 (223) | 682 (345)
HIV Viral Load of <20 detectable copies of HIV viral load [Count of Participants; unit: Participants] | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Methicillin-resistant Staphylococcus Aureus (MRSA) Colonization
Description: Participants were decolonized with a standard Methicillin-resistant Staphylococcus aureus (MRSA) decolonization protocol and monitored for 6 months. This is the number of participants who screened positive for Methicillin-resistant Staphylococcus aureus (MRSA) 6 months after being decolonized (i.e., recurrent infection)
Time Frame: 6 months
Population: Only participants who received the decolonization protocol and completed the 6 month follow-up visit (7 for "individual alone' and 6 for 'Individual plus household') were included in the analysis. The rest were lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Alone | Individual Plus Household
Number analyzed (Participants) | 7 | 6
Participants | 2 | 3
Statistical Analysis 1: Comparison: Individual Alone vs Individual Plus Household; Due to low enrollment in the intervention, statistical analysis was not possible; Test type: Other — The study was powered for enrollment of 100 subjects with MRSA colonization at baseline. Despite substantial screening, we were unable to enroll enough subjects to meet the necessary sample size; The study was powered for enrollment of 100 subjects with MRSA colonization at baseline. Despite substantial screening, we were unable to enroll enough subjects to meet the necessary sample size

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Individual Alone | Individual Plus Household
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Alone (N=9) | Individual Plus Household (N=9)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2014-08-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02029872/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2013-06-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT02029872/Prot_SAP_001.pdf